CLINICAL TRIAL: NCT05339880
Title: Evaluation of Correlation Between Laryngospasm, Emergence Agitation and Oculocardiac Reflex in Strabismus Surgery
Brief Title: Relation Between Oculocardiac Reflex and Laryngospasm
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Adnan Bayram, Professor, TC Erciyes University
Other Study IDs: 2020/107
Record Dates: First submitted 2022-02-10; First posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-02

CONDITIONS: Eye Abnormalities; Arrythmia
Keywords: strabismus surgery; laryngospasm; oculocardiac reflex; emergence agitation
MeSH Terms: conditions — Eye Abnormalities; Arrhythmias, Cardiac; Laryngismus; Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate whether there is a significant relation between various arrhythmias during the surgeon's stretching the eye muscles and laryngospasm and emergence agitation in strabismus surgeries

DETAILED DESCRIPTION:
Background: Laryngospasm is one of the serious complications that can be seen in perioperative period, especially during anesthesia induction and extubation. The aim of this study is to evaluate whether there is a significant relation between various arrhythmias during the surgeon's stretching the eye muscles and laryngospasm and emergence agitation in strabismus surgeries

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for the strabismus surgery
* ASA 1-2 patients
* 2-65 yo patients

Exclusion Criteria:

* Patients with kidney, cardiac diseases
* Being treated with sedative or anticonvulsant drugs
* ASA 3-4 patients
* Patients with upper respiratory tract disease in the last 2 weeks
* Patients who do not want to participate in the study
* Patients with behavioral disorders

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric and adult patients whose ages ranged between 2-18 and 18-65 and from the group of American Society of Anesthesiology (ASA) I-II who will have elective strabismus surgery
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-05-15 (Estimated); Study Completion 2022-05-15 (Estimated)

PRIMARY OUTCOMES:
Laryngospasm ratio | an average of 20 minutes during emergence
  Laryngospasm during emergence in patients with oculocardiac reflex in surgery will be recorded

SECONDARY OUTCOMES:
Emergence agitation in children | an average of 30 minutes
  The Paediatric Anaesthesia Emergence Delirium(PAED) score/scale will be evaluated. There are five scale items in PAED scale. Each item is scored from 1 to 4 and the scores are summed to obtain a total scale score. Higher scores indicate emergence agitation in the patient.
Emergence agitation in adults | an average of 30 minutes
  Aono's Four Point Agitation Scale will be evaluated. There are four scores from 1 to 4 on the scale. A high score is associated with emergence agitation in the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Bayram, Professor, Study Director — TC Erciyes University; Ahmet Cakir, MD, Principal Investigator — TC Erciyes University
Locations (1):
- Erciyes University, Kayseri, Melikgazi, Turkey (Türkiye)